CLINICAL TRIAL: NCT01301872
Title: Effect of Mechanical Ventilation Strategy on Lung Injury in Patients With Less Severe Acute Respiratory Distress Syndrome: Targeted on RAGE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 201012005RB
Record Dates: First submitted 2011-02-18; First posted 2011-02-23 (Estimated); Last update posted 2012-12-27 (Estimated); Status verified 2012-11

CONDITIONS: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): All patients meet ALI/less severe ARDS criteria
  Interventions: Other: check biomarker :RAGE

INTERVENTIONS:
Other: check biomarker :RAGE — We will check RAGE for all patients who have ARDS included in our study

SUMMARY:
During the past two decades, there current concept has evolved significantly that ventilator-induced lung injury (VILI) may not only impose a direct mechanical stress and subsequent injury to the lungs, but may also induce local as well as systemic inflammation responses, generally referred as biotrauma.1 Patients with ARDS often die of severe systemic inflammatory response syndrome (SIRS) and multiorgan dysfunction2 rather than refractory hypoxemia. Ranieri et al found that patients with less severe ARDS, i.e., a lung injury score of 2.5 or less, receiving ventilation with lung protective strategy involving low tidal volume (7.5 mL/kg PBW) and high PEEP could attenuate the pulmonary and systemic cytokine response compared with conventional ventilation with high tidal volume.3 Stuber et al found an increase in pro-inflammatory cytokines in the lung and plasma of patients with ARDS within 1 hour after switching the patients from a protective to non-protective ventilator strategy.4 The receptor for advanced glycation end-products (RAGE) was recently identified as a marker of injury to the alveolar type I epithelial cells5. Clinical studies showed that the plasma level of RAGE was associated with severity of lung injury and clinical outcome, and low tidal volume strategy ventilation accelerated the decline in plasma RAGE levels. These results suggest plasma RAGE level might be a reliable biomarker of alveolar epithelial injury in acute lung injury and may associated with ventilator induced lung injury6. Although, current approach to mechanical ventilation of a patient with ARDS emphasizes the use of lower tidal volumes with lower plateau pressures to avoid causing lung overdistension and ventilator associated lung injury (VILI)7; however, in the real world, some studies showed that strictly reduction of tidal volume to 6ml/kg PBW was modest in modern time, and was noticed only in patients with greater lung injury scores8. The benefit of VT strictly reduction to 6ml/kgPBW and its effect on VILI in patients with less severe ARDS whose Pplat are already below 30 cmH2O are controversy9. One of the possible solutions is to look at the biomarkers of injury to alveolar epithelial cells. Of these potentially promising markers, the receptor for advanced glycation end-product (RAGE) is of great interest.

We hypothesize that a strategy with strict low tidal volume in less severe ARDS and ALI patients with good compliance may be beneficial to this patient population. Therefore, we wish to propose a prospective single-center study to investigate the effect of mechanical ventilation strategy on the plasma level of RAGE in patients with less severe ARDS and acute lung injury.

DETAILED DESCRIPTION:
During the past two decades, there current concept has evolved significantly that ventilator-induced lung injury (VILI) may not only impose a direct mechanical stress and subsequent injury to the lungs, but may also induce local as well as systemic inflammation responses, generally referred as biotrauma.1 Patients with ARDS often die of severe systemic inflammatory response syndrome (SIRS) and multiorgan dysfunction2 rather than refractory hypoxemia. Ranieri et al found that patients with less severe ARDS, i.e., a lung injury score of 2.5 or less, receiving ventilation with lung protective strategy involving low tidal volume (7.5 mL/kg PBW) and high PEEP could attenuate the pulmonary and systemic cytokine response compared with conventional ventilation with high tidal volume.3 Stuber et al found an increase in pro-inflammatory cytokines in the lung and plasma of patients with ARDS within 1 hour after switching the patients from a protective to non-protective ventilator strategy.4 The receptor for advanced glycation end-products (RAGE) was recently identified as a marker of injury to the alveolar type I epithelial cells5. Clinical studies showed that the plasma level of RAGE was associated with severity of lung injury and clinical outcome, and low tidal volume strategy ventilation accelerated the decline in plasma RAGE levels. These results suggest plasma RAGE level might be a reliable biomarker of alveolar epithelial injury in acute lung injury and may associated with ventilator induced lung injury6. Although, current approach to mechanical ventilation of a patient with ARDS emphasizes the use of lower tidal volumes with lower plateau pressures to avoid causing lung overdistension and ventilator associated lung injury (VILI)7; however, in the real world, some studies showed that strictly reduction of tidal volume to 6ml/kg PBW was modest in modern time, and was noticed only in patients with greater lung injury scores8. The benefit of VT strictly reduction to 6ml/kgPBW and its effect on VILI in patients with less severe ARDS whose Pplat are already below 30 cmH2O are controversy9. One of the possible solutions is to look at the biomarkers of injury to alveolar epithelial cells. Of these potentially promising markers, the receptor for advanced glycation end-product (RAGE) is of great interest.

We hypothesize that a strategy with strict low tidal volume in less severe ARDS and ALI patients with good compliance may be beneficial to this patient population. Therefore, we will to propose a prospective single-center study to investigate the effect of mechanical ventilation strategy on the plasma level of RAGE in patients with less severe ARDS and acute lung injury.

ELIGIBILITY:
Inclusion Criteria:

* All intubated and mechanically ventilated patients who meet the criteria of American-European Consensus Conference (AECC) criteria for ALI/ ARDS:

Acute onset of illness Bilateral (patchy, diffuse, or homogeneous) infiltrates consistent with pulmonary edema PaO2/FiO2 <= 300 (corrected for altitude): (P/F <300 for ALI and P/F <200 for ARDS) No clinical evidence of left atrial hypertension

Exclusion Criteria:

* 1. Age <18 years 2. Enrolled in other clinical trials 3. Had confirmed alternative diagnoses that would have different clinical course than ARDS/ALI, e.g., diffuse alveolar hemorrhage, vasculitis, interstitial pneumonitis, etc.

  4. Congestive heart failure related pulmonary edema 5. Acute myocardial infarction 6. Pregnancy 7. Patients with definite contraindication to the use of low-tidal volume ventilation, e.g., increased intracranial pressure, tricyclic antidepressant overdose, etc.

  8. The patient who meets inclusion criteria initially but rapidly improved within 24 hours of diagnosis of ARDS/ALI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
the effect of mechanical ventilation strategy on the plasma level of RAGE in patients with less severe ARDS and acute lung injury. | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Jih-Shuin Jerng, MD,PhD, Principal Investigator — National Taiwan University Hospital